CLINICAL TRIAL: NCT01720927
Title: Pakistan Epidemiological Survey in Acute Pharyngitis
Status: Completed | Type: Observational
Sponsor: Suresh Kumar (Other)
Collaborators: Isra University (Other)
Responsible Party: Sponsor-Investigator, Suresh Kumar, Investigator, Hill Park General Hospital
Organization: Hill Park General Hospital (Other)
Other Study IDs: PK-12-02
Record Dates: First submitted 2012-11-01; First posted 2012-11-02 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Acute Pharyngitis
Keywords: Acute Pharyngitis, GABHS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Pharyngitis: Subjects presenting with acute pharyngitis

SUMMARY:
GABHS are common etiological agents for acute pharyngitis. However, local data is limited and large scale surveillance studies have not been done. This study aims to evaluate the disease burden in the community due to GABHS.

In this study, patients presenting with signs of acute pharyngitis will be evaluated. Patients with fulfilling the inclusion criteria will be tested for Rapid Antigen Detection test (RADT)

DETAILED DESCRIPTION:
Pharyngitis is a common reason for patients' visit to doctors. Group A beta- hemolytic streptococci (GABHS) account for 15-30 percent of cases of acute pharyngitis in children and 5 to 20 percent in adults1.

Because the signs and symptoms of GABHS pharyngitis overlap extensively with other infectious causes, making a diagnosis based solely on clinical findings is difficult. In patients with acute febrile respiratory illness, physicians accurately differentiate bacterial from viral infections using only the history and physical findings about one half of the time.2 No single element of the patient's history or physical examination reliably confirms or excludes GABHS pharyngitis.3 Sore throat, fever with sudden onset (temperature greater than 100.4° F [38° C]), and exposure to Streptococcus within the preceding two weeks suggest GABHS infection. Cervical node lymphadenopathy and pharyngeal or tonsillar inflammation or exudates are common signs. Palatal petechiae and scarlatiniform rash are highly specific but uncommon; a swollen uvula is sometimes noted. Cough, coryza, conjunctivitis, and diarrhea are more common with viral pharyngitis.

The original Centor score uses four signs and symptoms to estimate the probability of acute streptococcal pharyngitis in adults with a sore throat.4 The score was later modified by adding age and validated in 600 adults and children.5,6 The cumulative score determines the likelihood of streptococcal pharyngitis.

Rapid Antigen Detection Tests (RADTs) have been developed for the identification of GABHS directly from throat swabs. Although these rapid tests are more expensive than blood agar culture, they provide results faster. Rapid identification and treatment of patients with streptococcal pharyngitis can reduce the risk of the spread of group A b-hemolytic streptococci, allowing the patient to return to school or work sooner, and can reduce the acute morbidity associated with the illness. The use of RADTs for certain populations (e.g., patients in emergency departments) has been shown to significantly increase the number of patients who are appropriately treated for streptococcal pharyngitis, compared with use of traditional throat cultures.7

The great majority of the RADTs that are currently available have an excellent specificity of 95%, compared with blood agar plate culture. This means that false-positive test results are unusual, and, therefore, therapeutic decisions can be made with confidence on the basis of a positive test result. Unfortunately, the sensitivity of most of these tests is 80%-90%, or even lower, compared with blood agar plate culture. It has been suggested that most of the false-negative RADT results occur for patients who are merely Streptococcus carriers and are not truly infected. However, early studies of first-generation RADTs demonstrated that a large proportion of patients with false-negative RADT results were truly infected with group A b-hemolytic streptococci and were not merely carriers.8

Acute pharyngitis is commonly encountered in clinics and hospitals across Pakistan. It is common not only in children but also among adults. Limited data are available on the prevalence of this condition and existing data are from small single center based studies.

The available data from Pakistan suggest that the most common bacterial organism is GABHS, however, majority of throat swabs did not yield any isolate.9 The signs and symptoms of GABHS pharyngitis overlap extensively with other infectious causes, thus to make an etiologic diagnosis based solely on clinical findings is difficult. Improving diagnosis of bacterial causes of pharyngitis will lead to more rational use of antibiotics among clinicians, and potentially have a positive impact on the development of bacterial resistance in community acquired infections.

The modified Centor score is a valid tool to estimate the probability of acute streptococcal pharyngitis in patients with a sore throat. (reference) Patients with a score of zero or 1 are at very low risk for streptococcal pharyngitis and do not require testing (i.e., throat culture or rapid antigen detection testing [RADT]) or antibiotic therapy. Patients with a score of 2 or 3 should be tested using RADT or throat culture; positive results warrant antibiotic therapy. Patients with a score of 4 or higher are at high risk of streptococcal pharyngitis, and empiric treatment may be considered. (reference)

RADT allows for earlier treatment, symptom improvement, and reduced disease spread.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with signs of acute pharyngitis (duration of symptoms < 14 days)
* Subjects with sore throat
* Fever with sudden onset (temperature > 100 0 F (380 C)
* Exposure to Streptococcus within the preceding 2 weeks
* Children 3 years of age and above
* Subjects / guardians giving written authorization to participate in the study

Exclusion Criteria:

* Recurrent or persistent cases of sore throat
* Complicated pharyngitis (peritonsillar abscesses, Lemierre disease, Vincent's angina)
* Severe comorbidity
* Immunosuppression or history of acute rheumatic fever
* Special circumstances, such as sore throat after travel in past 2 weeks, sore throat linked to sexual transmission or rare epidemics (e.g. diphtheria)

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include children and adults presenting with sore throat, temperature greater than 100.40 F, tonsillar exudates and cervical adenopathy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 5140 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of GABHS in patients with acute pharyngitis. | 12 months

SECONDARY OUTCOMES:
To study the prevalence of GABHS in acute pharyngitis across different age groups. | 12 months
To study the correlation of centor score and RADT results. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- ISRA University, Hyderābād, Sindh, Pakistan